CLINICAL TRIAL: NCT01006824
Title: Randomized Controlled Trial of Wireless Capsule Endoscopy in the Evaluation of Obscure Gastrointestinal Bleeding
Brief Title: Trial of Wireless Capsule Endoscopy in the Evaluation of Obscure Gastrointestinal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Loren Laine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-02C010
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Obscure Gastrointestinal Bleeding (Occult or Overt)
Keywords: Capsule endoscopy; gastrointestinal hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Capsule Endoscopy
  Interventions: Other: Capsule endoscopy
- 2 (Active Comparator): Dedicated small bowel contrast radiography
  Interventions: Other: Dedicated small bowel contrast radiography

INTERVENTIONS:
Other: Capsule endoscopy — Capsule endoscopy
  Arms: 1
Other: Dedicated small bowel contrast radiography — Dedicated small bowel contrast radiography
  Arms: 2

SUMMARY:
This study compares wireless capsule endoscopy (patients swallow a pill-size camera that sends pictures of the intestine to a recorder worn on their belt) to an x-ray study (called dedicated small bowel contrast radiography) in patients who have bleeding from the gastrointestinal tract without a source of the bleeding identified on routine endoscopic examinations of the esophagus (food pipe), stomach, small intestine, and large intestine.

The investigators hope to determine if the capsule is a better test in terms of decreasing further bleeding, decreasing the need for further diagnostic testing, and decreasing the need for blood transfusions and time spent in the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Iron deficiency anemia in men or post-menopausal women and positive fecal occult blood test in pre-menopausal women with nondiagnostic upper endoscopy, colonoscopy, and push enteroscopy.
2. Persistent or recurrent melena or hematochezia with nondiagnostic upper endoscopy, colonoscopy, and push enteroscopy.

Exclusion Criteria:

1. Known or suspected GI tract obstruction
2. Severe motility disorders (e.g., achalasia, gastroparesis, pseudoobstruction)
3. Pregnancy
4. Cardiac pacemaker or implanted electro-medical devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2003-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Further bleeding | 1 year

SECONDARY OUTCOMES:
Diagnostic yield | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, M.D., Principal Investigator — University of Southern California
Locations (1):
- L.A. County + U.S.C. Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Laine L, Sahota A, Shah A. Does capsule endoscopy improve outcomes in obscure gastrointestinal bleeding? Randomized trial versus dedicated small bowel radiography. Gastroenterology. 2010 May;138(5):1673-1680.e1; quiz e11-2. doi: 10.1053/j.gastro.2010.01.047. Epub 2010 Feb 2. PMID 20138043